CLINICAL TRIAL: NCT06336369
Title: BiliMetHealth- Energy Metabolism and Brown Adipose Tissue (BAT) Activity in Individuals With Gilbert's Syndrome (GS) and Healthy Controls
Brief Title: Brown Adipose Tissue Activity in Gilbert's Syndrome
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: University of Vienna (Other); Griffith University (Other)
Responsible Party: Principal Investigator, Dr. Florian Kiefer, Florian Kiefer MD, PhD, Medical University of Vienna
Other Study IDs: 1713/2023
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Gilbert Syndrome
MeSH Terms: conditions — Gilbert Disease | interventions — Body Composition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Cases: (Gilbert-Syndrom):
  * Total bilirubin in the blood > 1.2 mg/dL (17.1 μM)
  * Unconjugated (indirect bilirubin) > 1 mg/dL
  Interventions: Diagnostic Test: analyzing brown adipose tissue, body composition and metabolic health
- Controls: Controls (non-Gilbert-Syndrom):
  * Total bilirubin in the blood ≤ 1.2 mg/dL (17.1 μM)
  * Unconjugated (indirect bilirubin) ≤ 1 mg/dL
  Interventions: Diagnostic Test: analyzing brown adipose tissue, body composition and metabolic health

INTERVENTIONS:
Diagnostic Test: analyzing brown adipose tissue, body composition and metabolic health — cooling procedure, PET-CT imaging, MR imaging, blood sampling, indirect calorimetry, thermograpy, impedance analysis

SUMMARY:
The goal of this case-control study is to investigate energy metabolism and brown adipose tissue (BAT) activity in individuals with Gilbert's syndrome (GS) and controls. The main focus of the study is to analyze:

1. the link between bilirubin metabolism and metabolic health.
2. energy metabolism and body composition in individuals with Gilbert's syndrome and control subjects
3. brown adipose tissue activity in Gilbert's syndrome and healthy controls.

Participants will undergo the following investigations:

1. cold exposure
2. PET-CT imaging with 18-F-FDG
3. MRI imaging of liver, abdominal fat and muscle
4. blood sampling
5. indirect calorimetry
6. bioelectrical impedance analysis
7. infrared thermography

Researchers will compare individuals with GS and control subjects in terms of metabolic health, body composition and BAT activity.

DETAILED DESCRIPTION:
Bilirubin has long been associated with liver pathology and haemolytic conditions and was until recently assumed to possess little or no biological function. However, unconjugated bilirubin (UCB) rarely approaches these toxic levels and approximates 10 μM in the general population, which is 30-60 times below the reported toxic threshold.

The beneficial associations of mildly elevated blood UCB concentrations with diseases of civilization (in particular those affecting the cardiovascular system and all-cause mortality) have been reported in numerous studies. In addition, a mildly elevated UCB is also associated with reduced adiposity, decreased risk of metabolic syndrome, non-alcoholic fatty liver disease and diabetes as well as overall cancer risk. Bilirubin downregulates pro-inflammatory responses often observed in disease, which complements epidemiological evidence of reduced inflammatory, autoimmune, and degenerative diseases in individuals with GS. Together, these observations may account for the reduced all-cause mortality rates reported in those with GS compared to the normobilirubinaemic population. Finally, bilirubin has been recently reported to modulate cell signalling and act as an endocrine molecule. We were amongst the first to show that - bile pigments possess substantial anti-mutagenic in vitro and ex vivo antioxidant capacity; - subjects with mild hyperbilirubinaemia - also called Gilbert ́s Syndrome (GS) have a significantly reduced BMI compared to age and gender matched controls, a lower hip circumference (HC) as well as lower total/LDL cholesterol, triglycerides and low- and pro-atherogenic sub fractions as well as IL-6. Interestingly effects of GS in older participants (≥35yrs) is most profound, with substantially reduced anthropometric data and improved lipid profile.

Very recently we and others showed that enhanced lipid catabolism in GS seems to be the key mechanism involved.

Based on these very preliminary observations, and the strong link between bilirubin metabolism and metabolic health we aim to investigate in this application more deeply mechanistic questions to better understand why GS subjects show the very specific phenotype and its metabolic potential.

Here we propose a human case control study. Therefore we will investigate 40 GS individuals vs. 40 age and gender matched controls. Participants will be recruited as performed in previous studies.

Cases: (Gilbert-Syndrom):

* Total bilirubin in the blood > 1.2 mg/dL (17.1 μM)
* Unconjugated (indirect bilirubin) > 1 mg/dL

Controls (non-Gilbert-Syndrom):

* Total bilirubin in the blood ≤ 1.2 mg/dL (17.1 μM)
* Unconjugated (indirect bilirubin) ≤ 1 mg/dL

The duration of the study lasts for every participant 3 independent days. On the preinvestigation-day a screening will be performed including a blood sampling to prove in- and exclusion criteria.

On study day 1 participants must be fastened and will undergo the measurement of the brown adipose tissue.

On study day 2 participants must be fastened and will undergo the measurement of fat distribution in liver and muscle.

One 24-hr recall, a FFQ and a physical activity questionnaire will be assessed at the beginning of study day 1.

ELIGIBILITY:
Inclusion Criteria:

* written consent, age between 18 and 65 years of age, liver marker (AST, ALT, GGT) < 2x of the upper norm range, non-smoker, moderate physical activity, ability to understand the requirements of the course of study

Cases: (Gilbert-Syndrom):

* Total bilirubin in the blood > 1.2 mg/dL (17.1 μM)
* Unconjugated (indirect bilirubin) > 1 mg/dL

Controls (non-Gilbert-Syndrom):

* Total bilirubin in the blood ≤ 1.2 mg/dL (17.1 μM)
* Unconjugated (indirect bilirubin) ≤ 1 mg/dL

Exclusion Criteria:

* age < 18 or > 65 years; having current or any history of cardio-pulmonary, metabolic or musculoskeletal disease; breastfeeding or was/potentially pregnant; liver diseases incl. hep A and B; kidney diseases; active tumor disease; persons with an organ transplant; not willing to meet the demands of the study; not being weight stable (± 5% body mass; self-reported) for at least the 3 months prior to their involvement; or any conditions or concurrent behaviour (including medication) that may have posed undue personal risk to the participant, introduce bias to the study or were influencing liver marker in the last 5 weeks.

Cases: (Gilbert-Syndrom):

* Total bilirubin in the blood ≤ 1.2 mg/dL (17.1 μM)
* Unconjugated (indirect bilirubin) ≤ 1 mg/dL

Controls (non-Gilbert-Syndrom):

* Total bilirubin in the blood > 1.2 mg/dL (17.1 μM)
* Unconjugated (indirect bilirubin) > 1 mg/dL

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: cohort from previous study
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
cold-induced brown adipose tissue (BAT) activation | 3 independent days, 12 hours in total
  proven via PET-CT imaging due to radioactive tracer uptake (18-F-FDG)

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Heinz Wagner, Univ.-Prof. Mag., Principal Investigator — University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bulmer AC, Blanchfield JT, Toth I, Fassett RG, Coombes JS. Improved resistance to serum oxidation in Gilbert's syndrome: a mechanism for cardiovascular protection. Atherosclerosis. 2008 Aug;199(2):390-6. doi: 10.1016/j.atherosclerosis.2007.11.022. Epub 2007 Dec 26. PMID 18155709
- [Background] Wagner KH, Wallner M, Molzer C, Gazzin S, Bulmer AC, Tiribelli C, Vitek L. Looking to the horizon: the role of bilirubin in the development and prevention of age-related chronic diseases. Clin Sci (Lond). 2015 Jul;129(1):1-25. doi: 10.1042/CS20140566. PMID 25881719
- [Background] Wagner KH, Shiels RG, Lang CA, Seyed Khoei N, Bulmer AC. Diagnostic criteria and contributors to Gilbert's syndrome. Crit Rev Clin Lab Sci. 2018 Mar;55(2):129-139. doi: 10.1080/10408363.2018.1428526. Epub 2018 Feb 1. PMID 29390925
- [Background] Vitek L. The role of bilirubin in diabetes, metabolic syndrome, and cardiovascular diseases. Front Pharmacol. 2012 Apr 3;3:55. doi: 10.3389/fphar.2012.00055. eCollection 2012. PMID 22493581
- [Background] Vitek L. Bilirubin and atherosclerotic diseases. Physiol Res. 2017 Apr 5;66(Suppl 1):S11-S20. doi: 10.33549/physiolres.933581. PMID 28379026
- [Background] Weaver L, Hamoud AR, Stec DE, Hinds TD Jr. Biliverdin reductase and bilirubin in hepatic disease. Am J Physiol Gastrointest Liver Physiol. 2018 Jun 1;314(6):G668-G676. doi: 10.1152/ajpgi.00026.2018. Epub 2018 Mar 1. PMID 29494209
- [Background] Jangi S, Otterbein L, Robson S. The molecular basis for the immunomodulatory activities of unconjugated bilirubin. Int J Biochem Cell Biol. 2013 Dec;45(12):2843-51. doi: 10.1016/j.biocel.2013.09.014. Epub 2013 Oct 19. PMID 24144577
- [Background] Horsfall LJ, Nazareth I, Pereira SP, Petersen I. Gilbert's syndrome and the risk of death: a population-based cohort study. J Gastroenterol Hepatol. 2013 Oct;28(10):1643-7. doi: 10.1111/jgh.12279. PMID 23701650
- [Background] Vitek L, Haluzik M. The role of bile acids in metabolic regulation. J Endocrinol. 2016 Mar;228(3):R85-96. doi: 10.1530/JOE-15-0469. Epub 2016 Jan 5. PMID 26733603
- [Background] Bulmer AC, Ried K, Blanchfield JT, Wagner KH. The anti-mutagenic properties of bile pigments. Mutat Res. 2008 Jan-Feb;658(1-2):28-41. doi: 10.1016/j.mrrev.2007.05.001. Epub 2007 May 18. PMID 17602853
- [Background] Bulmer AC, Ried K, Coombes JS, Blanchfield JT, Toth I, Wagner KH. The anti-mutagenic and antioxidant effects of bile pigments in the Ames Salmonella test. Mutat Res. 2007 May 18;629(2):122-32. doi: 10.1016/j.mrgentox.2007.01.008. Epub 2007 Feb 11. PMID 17350329
- [Background] Wallner M, Blassnigg SM, Marisch K, Pappenheim MT, Mullner E, Molzer C, Nersesyan A, Marculescu R, Doberer D, Knasmuller S, Bulmer AC, Wagner KH. Effects of unconjugated bilirubin on chromosomal damage in individuals with Gilbert's syndrome measured with the micronucleus cytome assay. Mutagenesis. 2012 Nov;27(6):731-5. doi: 10.1093/mutage/ges039. Epub 2012 Aug 8. PMID 22874647
- [Background] Wallner M, Antl N, Rittmannsberger B, Schreidl S, Najafi K, Mullner E, Molzer C, Ferk F, Knasmuller S, Marculescu R, Doberer D, Poulsen HE, Vitek L, Bulmer AC, Wagner KH. Anti-genotoxic potential of bilirubin in vivo: damage to DNA in hyperbilirubinemic human and animal models. Cancer Prev Res (Phila). 2013 Oct;6(10):1056-63. doi: 10.1158/1940-6207.CAPR-13-0125. Epub 2013 Aug 27. PMID 23983086
- [Background] Seyed Khoei N, Grindel A, Wallner M, Molzer C, Doberer D, Marculescu R, Bulmer A, Wagner KH. Mild hyperbilirubinaemia as an endogenous mitigator of overweight and obesity: Implications for improved metabolic health. Atherosclerosis. 2018 Feb;269:306-311. doi: 10.1016/j.atherosclerosis.2017.12.021. Epub 2017 Dec 14. PMID 29279144
- [Background] Wallner M, Marculescu R, Doberer D, Wolzt M, Wagner O, Vitek L, Bulmer AC, Wagner KH. Protection from age-related increase in lipid biomarkers and inflammation contributes to cardiovascular protection in Gilbert's syndrome. Clin Sci (Lond). 2013 Sep;125(5):257-64. doi: 10.1042/CS20120661. PMID 23566065
- [Background] Molzer C, Wallner M, Kern C, Tosevska A, Schwarz U, Zadnikar R, Doberer D, Marculescu R, Wagner KH. Features of an altered AMPK metabolic pathway in Gilbert's Syndrome, and its role in metabolic health. Sci Rep. 2016 Jul 21;6:30051. doi: 10.1038/srep30051. PMID 27444220
- [Background] Stec DE, John K, Trabbic CJ, Luniwal A, Hankins MW, Baum J, Hinds TD Jr. Bilirubin Binding to PPARalpha Inhibits Lipid Accumulation. PLoS One. 2016 Apr 12;11(4):e0153427. doi: 10.1371/journal.pone.0153427. eCollection 2016. PMID 27071062
- [Background] Hana CA, Tran LV, Molzer C, Mullner E, Hormann-Wallner M, Franzke B, Tosevska A, Zohrer PA, Doberer D, Marculescu R, Bulmer AC, Freisling H, Moazzami AA, Wagner KH. Serum metabolomics analysis reveals increased lipid catabolism in mildly hyperbilirubinemic Gilbert's syndrome individuals. Metabolism. 2021 Dec;125:154913. doi: 10.1016/j.metabol.2021.154913. Epub 2021 Oct 20. PMID 34653509